CLINICAL TRIAL: NCT02939859
Title: Use of Cellular Stromal Vascular Fraction (cSVF) for Select Multiple Sclerosis, Autoimmune, Inflammatory, and Neurologic Conditions: Clinical Interventional Study of Adverse Events and Clinical Outcomes Using Autologous Stem-Stromal Cells.
Brief Title: Use of Cellular Stromal Vascular Fraction in Multiple Sclerosis,Autoimmune, Inflammatory, Neurologic Conditions
Acronym: cSVF
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawn [COVID restrictions prevent patient enrollment or treatment. Clinical Trial facility is being closed due to viral limitations and loss of staff to perform]
Sponsor: Healeon Medical Inc (Industry)
Collaborators: Global Alliance for Regenerative Medicine (Other)
Responsible Party: Principal Investigator, Robert W. Alexander, MD, FICS, Principal Investigator, Science, Healeon Medical Inc
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGV-GARM
Record Dates: First submitted 2016-10-03; First posted 2016-10-20 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Multiple Sclerosis; Autoimmune
Keywords: Multiple Sclerosis; Demyelinating Diseases; Nervous System Diseases; Autoimmune Disorders
MeSH Terms: conditions — Multiple Sclerosis; Demyelinating Diseases; Nervous System Diseases; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Microcannula Harvest Adipose (Experimental): Acquisition AD-tSVF via closed syringe microcannula
  Interventions: Procedure: Microcannula Harvest Adipose
- Centricyte 1000 (Experimental): Autologous Adipose-Derived Tissue Stromal Vascular Fraction (AD-tSVF) via enzymatic isolation/concentration via Centricyte 1000 Closed System to create AD-cSVF
  Interventions: Device: Centricyte 1000
- Sterile Normal Saline (Experimental): Re-suspension of Autologous AD-cSVF pellet in Normal Saline deployment via IV
  Interventions: Procedure: Sterile Normal Saline IV deployment AD-cSVF

INTERVENTIONS:
Procedure: Microcannula Harvest Adipose — Use of Closed Syringe Microcannula Harvest Autologous Adipose-Derived Stem/Stromal Cells
  Arms: Microcannula Harvest Adipose
Device: Centricyte 1000 — Use of Centricyte 1000 closed system digestion adipose tissue stromal vascular fraction to create a AD-cSVF
  Arms: Centricyte 1000
Procedure: Sterile Normal Saline IV deployment AD-cSVF — Sterile Normal Saline Suspension AD-cSVF in 500 cc IV use
  Arms: Sterile Normal Saline

SUMMARY:
Purpose of study is to determine safety and efficacy of use of autologous Adipose-Derived cellular Stromal Vascular Fraction (AD-cSVF) suspended in Normal Saline and delivered via intravascular system of quality of life and alteration of documented Muscular Sclerosis (MS) and related neurodegenerative patients. It is believed that the heterogeneous cell population which includes multipotent stem/stromal cells are capable of immune modulation/inflammatory modulation properties. Exam of disease progression and quality of life changes will be evaluated.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a demyelination disease which features damage to insulating covers of nerve cells in the brain and spinal cord. This damage or degenerative changes disrupts the ability of parts of the nervous system to communicate, resulting in range of signs and symptoms which include physical and mental changes.

Symptoms are variable and often include visual changes, sensory irregularities, and motor coordination. MS has several forms which result in new symptoms in either isolated attacks (relapsing forms) or gradual increasing symptoms (progressive forms).

While cause is not clear, mechanisms have been suggested association with loss of the immune system or failure to produce myelin-producing cells. Some suggest a genetic predisposition or environmental factor, but the exact causation in all cases have not been elucidated.

Medications have been developed, but remain modestly effective and possessing major side effects and poorly tolerated. Alternative treatments, including physical therapy and some stem/stromal therapies have become more common.

Three main characteristics of MS are: 1). Lesion formations in the central nervous system (called Plaques); 2). Inflammation; 3). Destruction of myelin sheaths of neurons. This demyelination is thought to stimulate the inflammatory processes due to action of a lymphocyte group known at T-cell which seems to recognize patient's own myelin as foreign and proceeds to attack it (known as "autoreactive lymphocytes").

Traditionally, exacerbation's are often treated with high dose intravenous steroids which may be of short term reduction of symptoms, not addressing the underlying causation. Current medications available for treatment are expensive and fraught with major side effects, making their use very difficult and producing limited measured value.

With the advent of convenient adipose harvesting and processing in closed systems, the ability to easily and safely acquire significant of stem/stromal cells, studies are underway to utilize autologous stem/stromal cells. This study is aimed at evaluation of the safety profile (adverse reactions & severe adverse reaction) of the closed syringe, microcannula harvesting of subdermal fat deposits. This autologous cell group obtained with isolation and concentration of cells within the stromal vascular fraction (SVF) via enzymatic digestion, and deployed via intravascular routes. As these cells are very small, there is belief that they are able to pass into the cerebral fluids in defects of the blood brain barrier (BBB) or are small enough to pass into the fluids of the CNS (central nervous system).

ELIGIBILITY:
Inclusion Criteria:

* Documented functional damage to central or peripheral nervous system unlikely to improve with present standard of care
* At least 6 months after onset of disease process
* If under current medical therapy (drug or surgical) for the condition, patient considered stable on that treatment and unlikely to have significant reversal of associated neurological functions damage as a result of ongoing treatments
* In estimation of providers and neurologists have the potential for improvement with AD-cSVF treatment, and be at minimal risk of potential harm from the procedure
* Over 18 year old, and capable of providing informed consent
* Medically stable and cleared by primary care physician, neurologist, or licensed practitioner that patient is felt to be reasonably expected to be expected to undergo procedures without known significant risk to health

Exclusion Criteria:

* Patient must be capable of an adequate neurologic examination and evaluation to document the pathology and ability to cooperate with examination
* Patient much be capable and willing to undergo follow up neurologic exams with investigators or their own neurologists
* Patient must be capable and competent to provide informed consent to participation
* In estimation of investigators, the patient may be at increased or significant risk of harm to the patient's general health or neurologic functions for collection of AD-cSVF collection
* Patients not medically stable, or who may be at significant risk to their health undergoing any and all procedures will not be eligible
* Women of childbearing age must not be pregnant at the time of treatment, and should refrain from becoming pregnant for 3 months post-treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events [Time Frame: Outcome measures evaluated at baseline and reviewed at 6 month intervals for average time frame of 5 years] | 6 month intervals for up to 5 years
  Activities of Daily Living (ADL)

SECONDARY OUTCOMES:
Neurologic Functioning | 6 month intervals for up to 5 years
  Deficits of neurologic function identified by patient as impaired prior to treatment assessed. Examples: neurologic function may include speech, balance, motor/sensory actions, hearing, gait, strength, pain, paresthesias
Quality of Life Questionnairre | 1 year
  Change from baseline in overall General Quality of Life (GQL) Health status questionnaire (SF-36)
Fatigue | 6 month intervals for up to 5 years
  Change from baseline measured by modified fatigue impact scale (MFIS)
Cognitive Problems | 1 year intervals for up to 5 years
  Cognitive Problems measured by Perceived Deficits Questionnaire (PDQ)
Brain Lesions | 6 month intervals for up to 5 years
  PIXYL Software Analysis from Baseline and at 6 month MRI with/without contrast Brain

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Alexander, MD, Principal Investigator — GARM International; Glenn C Terry, MD, Principal Investigator — GARM
Locations (2):
- Regenevita LLC, Stevensville, Montana, United States
- Global Alliance for Regenerative Medicine (GARM), Roatán, Hn, Honduras

IPD SHARING:
Plan to Share IPD: Undecided
Annual Summary of Cases to All Collaborators

REFERENCES:
- [Background] Nakahara J, Maeda M, Aiso S, Suzuki N. Current concepts in multiple sclerosis: autoimmunity versus oligodendrogliopathy. Clin Rev Allergy Immunol. 2012 Feb;42(1):26-34. doi: 10.1007/s12016-011-8287-6. PMID 22189514
- [Background] Ascherio A, Munger KL. Environmental risk factors for multiple sclerosis. Part I: the role of infection. Ann Neurol. 2007 Apr;61(4):288-99. doi: 10.1002/ana.21117. PMID 17444504
- [Background] Tsang BK, Macdonell R. Multiple sclerosis- diagnosis, management and prognosis. Aust Fam Physician. 2011 Dec;40(12):948-55. PMID 22146321
- [Background] Huntley A. A review of the evidence for efficacy of complementary and alternative medicines in MS. Int MS J. 2006 Jan;13(1):5-12, 4. PMID 16420779
- [Background] Weinshenker BG. Natural history of multiple sclerosis. Ann Neurol. 1994;36 Suppl:S6-11. doi: 10.1002/ana.410360704. PMID 8017890
- [Background] Dyment DA, Ebers GC, Sadovnick AD. Genetics of multiple sclerosis. Lancet Neurol. 2004 Feb;3(2):104-10. doi: 10.1016/s1474-4422(03)00663-x. PMID 14747002
- [Background] Hassan-Smith G, Douglas MR. Epidemiology and diagnosis of multiple sclerosis. Br J Hosp Med (Lond). 2011 Oct;72(10):M146-51. doi: 10.12968/hmed.2011.72.sup10.m146. PMID 22041658
- [Background] Lublin FD, Reingold SC, Cohen JA, Cutter GR, Sorensen PS, Thompson AJ, Wolinsky JS, Balcer LJ, Banwell B, Barkhof F, Bebo B Jr, Calabresi PA, Clanet M, Comi G, Fox RJ, Freedman MS, Goodman AD, Inglese M, Kappos L, Kieseier BC, Lincoln JA, Lubetzki C, Miller AE, Montalban X, O'Connor PW, Petkau J, Pozzilli C, Rudick RA, Sormani MP, Stuve O, Waubant E, Polman CH. Defining the clinical course of multiple sclerosis: the 2013 revisions. Neurology. 2014 Jul 15;83(3):278-86. doi: 10.1212/WNL.0000000000000560. Epub 2014 May 28. PMID 24871874
- [Background] He D, Xu Z, Dong S, Zhang H, Zhou H, Wang L, Zhang S. Teriflunomide for multiple sclerosis. Cochrane Database Syst Rev. 2012 Dec 12;12:CD009882. doi: 10.1002/14651858.CD009882.pub2. PMID 23235682
- [Background] Manouchehrinia A, Constantinescu CS. Cost-effectiveness of disease-modifying therapies in multiple sclerosis. Curr Neurol Neurosci Rep. 2012 Oct;12(5):592-600. doi: 10.1007/s11910-012-0291-6. PMID 22782520
- [Background] Hassan-Smith G, Douglas MR. Management and prognosis of multiple sclerosis. Br J Hosp Med (Lond). 2011 Nov;72(11):M174-6. doi: 10.12968/hmed.2011.72.sup11.m174. PMID 22082979
- [Background] Freedman MS. Long-term follow-up of clinical trials of multiple sclerosis therapies. Neurology. 2011 Jan 4;76(1 Suppl 1):S26-34. doi: 10.1212/WNL.0b013e318205051d. PMID 21205679
- [Background] Bates D. Treatment effects of immunomodulatory therapies at different stages of multiple sclerosis in short-term trials. Neurology. 2011 Jan 4;76(1 Suppl 1):S14-25. doi: 10.1212/WNL.0b013e3182050388. PMID 21205678
- [Background] Martinelli Boneschi F, Vacchi L, Rovaris M, Capra R, Comi G. Mitoxantrone for multiple sclerosis. Cochrane Database Syst Rev. 2013 May 31;2013(5):CD002127. doi: 10.1002/14651858.CD002127.pub3. PMID 23728638
- [Background] Balak DM, Hengstman GJ, Cakmak A, Thio HB. Cutaneous adverse events associated with disease-modifying treatment in multiple sclerosis: a systematic review. Mult Scler. 2012 Dec;18(12):1705-17. doi: 10.1177/1352458512438239. Epub 2012 Feb 27. PMID 22371220
- [Background] Comi G. Treatment of multiple sclerosis: role of natalizumab. Neurol Sci. 2009 Oct;30 Suppl 2:S155-8. doi: 10.1007/s10072-009-0147-2. PMID 19882365
- [Background] Farinotti M, Vacchi L, Simi S, Di Pietrantonj C, Brait L, Filippini G. Dietary interventions for multiple sclerosis. Cochrane Database Syst Rev. 2012 Dec 12;12:CD004192. doi: 10.1002/14651858.CD004192.pub3. PMID 23235605
- [Background] Olsen SA. A review of complementary and alternative medicine (CAM) by people with multiple sclerosis. Occup Ther Int. 2009;16(1):57-70. doi: 10.1002/oti.266. PMID 19222053
- [Background] Miller AE. Multiple sclerosis: where will we be in 2020? Mt Sinai J Med. 2011 Mar-Apr;78(2):268-79. doi: 10.1002/msj.20242. PMID 21425270
- [Background] Luessi F, Siffrin V, Zipp F. Neurodegeneration in multiple sclerosis: novel treatment strategies. Expert Rev Neurother. 2012 Sep;12(9):1061-76; quiz 1077. doi: 10.1586/ern.12.59. PMID 23039386